CLINICAL TRIAL: NCT04541459
Title: Validation of New Devices Against Ambient Electromagnetic Radiation: A Randomized Double Blind Controlled Study
Brief Title: Validation of New Devices Against Ambient Electromagnetic Radiation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Waveguard GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: WAVEGUARD MALE FERTILITY CC01; IRB #20-329 (Other: Cleveland Clinic Institutional Review Board)
Record Dates: First submitted 2020-08-27; First posted 2020-09-09 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Intervention Model Description: Randomised double blind controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Qi-Shield user group (Sham Comparator)
  Interventions: Device: sham device against ambient electromagnetic radiation
- Qi-Shield user group (Active Comparator)
  Interventions: Device: new device against ambient electromagnetic radiation

INTERVENTIONS:
Device: new device against ambient electromagnetic radiation — New device provides protection against the radiations emitted by the smartphone and laptop devices. Device uses conductive fluids in a particular geometric arrangement intended to ameliorate the negative effects of EMW radiation.
  Arms: Qi-Shield user group
Device: sham device against ambient electromagnetic radiation — Sham device as as a control for new device, which provides protection against the radiations emitted by the smartphone and laptop devices. Device uses conductive fluids in a particular geometric arrangement intended to ameliorate the negative effects of EMW radiation.
  Arms: Sham Qi-Shield user group

SUMMARY:
Project Summary Cell phones have become indispensable devices in the investigator's daily life. These phones operate between 400 and 2000 MHz frequency bands and emit radiofrequency electromagnetic waves (EMW). Radio-frequency electro-magnetic field exposure from cell phones or other sources of microwaves have deleterious effects on sperm parameters (like sperm count, morphology, motility). Further, EMW radiation emitted by mobile phones affects cells and organelles, and results in disorientation of charged molecules within the cytosol and a distortion of electron flow along the internal membranes of the cells. These cellular changes results in the generation of ROS leading to oxidative stress, which in turn results in radiation-induced sperm DNA fragmentation.

Radiation shield can help provide protection from high levels of EMW radiations deflecting, diverting, and absorbing the radiation between the user and the source. A new EMW radiation shield, Qi-Shield device developed by Waveguard GmbH (Bautzen, Germany) provides protection against the radiations emitted by the smartphone and laptop devices. Qi-Shield utilizes conductive fluids in a particular geometric arrangement intended to ameliorate the negative effects of EMW radiation.

Study Aims:

To evaluate the changes in the semen parameters from the use of Qi-Shield device in sham (control) and user groups To determine the molecular changes pertaining to sperm proteins from the use of Qi-Shield device in sham (control) and user groups

Significance The negative health consequences of EMWs have been documented across a wide range of device types, exposure frequencies and doses (Giuliani, 2010), at field strengths substantially below the International Commission on Non-Ionizing Radiation Protection (ICNIRP) guidelines for permissible exposures. In the absence of a revision in the ICNIRP guidelines, near-term public exposures to EMWs will most certainly continue to increase, despite the scientific evidence suggesting more careful review and recommendations to limit exposure to electromagnetic fields as much as possible. At present, there is no veritable means for counteracting the negative health consequences of human-made EMWs, revealing an unmet need for a means of protecting from or ameliorating the negative effects of EMWs, and the need for devising strategies for creating safer living and working environments in a time of increasing EMW exposures.

Positive results in this study would demonstrate a means of counteracting negative effects on human sperm due to EMWs. Documentation of protection due to the Qi-Shield devices would show proof of principle that a low-cost passive device, portable and without battery or mains power, can provide improvements in human sperm parameters, with promise for a means of counteracting EMW-reduced fertility in large numbers of people. Confirmation of changes on protein expression would provide data needed to identify specific pathways of action, insight that is necessary for a more detailed understanding of the mechanisms of action of the EMW protection effect. Taken together, these results would suggest further lines of study in EMW protection, and provide clinical support for the adoption of EMW-protecting devices in the home and workplace.

DETAILED DESCRIPTION:
Normal healthy men enrolled in the study will be asked to provide semen specimens prior to the use of device. Samples will be produced with a minimum of 48-72 hours of abstinence. Further, the subjects will be blindly assigned with either sham Qi-Shield or Qi-Shield device and will be instructed to use the device for a duration of 8 weeks .Semen samples will be provided by the subjects at 0, 4 and 8 weeks interval.

Group 1 study subjects will be provided with sham Qi-Shield device, whereas Group 2 study subjects with be provided with actual Qi-Shield device. Each user will be provided with a small carrier bag to accommodate the device during their travel. The participants are advised to keep the device within 3 meters of range as per the manufacturer instructions for a duration of 8 weeks.

Semen analysis All specimens will be collected by masturbation at the Andrology Laboratory after 48-72 hours of sexual abstinence. Samples will be allowed to liquefy completely for 15-20 minutes at 37C before further processing. After complete liquefaction, semen analysis will be carried out using automated LensHooke™X1 PRO semen quality analyzer (Bonraybio Co., Ltd) to determine sperm concentration and motility, progressive motility (Agarwal et al., 2019). Viability will be determined by Eosin-Nigrosin stain if motility is <25%. Smears of the raw semen will be stained with a Diff-Quik kit (Baxter Healthcare Corporation, Inc., McGaw Park, IL) for assessment of sperm morphology according to strict criteria as described in the WHO, 5th edition guideline.

White blood cell measurement When the round cell concentration in the ejaculate is >1 X million/mL or >5 round cells per high power field, the sample will be tested for leukocytospermia, i.e. >1 X million white blood cells/mL. This will be confirmed by the peroxidase or the Endtz test.

Measurement of Oxidation Reduction Potential ORP measures the transfer of electrons from a reductant (or antioxidant) to an oxidant. ORP is measured in millivolts (mV). In the current study, ORP will be measured using novel galvanostat-based technology-the MiOXSYS System (Aytu Bioscience, Englewood, CO). Briefly, 30µL of liquefied semen will be loaded on the MiOXSYS sensor. The sensor will be inserted into the MiOXSYS analyzer. Static ORP (sORP), measured in mV, is the integrated measure of the existing balance between total oxidants and reductants in a biological system. Data will be normalized with sperm concentration. ORP will be expressed as mV/ million sperm/mL.

DNA fragmentation DNA fragmentation will be assessed via Terminal deoxynucleotidyl transferase-mediated dUTP nick-end labelling assay (TUNEL assay). Briefly, 2 million spermatozoa will be washed in phosphate buffered saline (PBS) and resuspended in 3.7% paraformaldehyde. A total of 2 aliquots (A and B) will be used for each donor, one for ORP measurement and other for measurement of sperm DNA fragmentation. These will be placed on ice for 30-60 minutes at 4C. Thereafter, the spermatozoa will again be washed to remove the paraformaldehyde and then re-suspended in 70% ice-cold ethanol, stored at -20C until the time of analysis.

Sperm DNA fragmentation will be evaluated using a TUNEL assay with an Apo-DirectTM kit (Pharmingen, San Diego, CA). Positive and negative kit controls provided by the manufacturer and positive test prepared by treating with hydrogen peroxide controls will be included for each run. Following a second wash in PBS to remove ethanol, the sperm pellets are re-suspended in 50 µL of freshly prepared staining solution for 60 minutes at 37C. The staining solution contains terminal deoxytransferase (TdT) enzyme, TdT reaction buffer, fluorescein isothiocynate tagged deoxyuridine triphosphate nucleotides (FITC-dUTP) and distilled water. All specimens are further washed in rinse buffer and re-suspended in 0.5 mL of propidium Iodide/RNase solution, and incubated for 30 minutes followed by flow cytometric analysis.

BD C6 Acuri cytometry analysis: All fluorescence signals of labelled spermatozoa will be analyzed by the flow cytometer BD Accuri Flow cytometer (Becton Dickinson, San Jose, CA). About 10,000 spermatozoa will be examined for each assay at a slow flow rate of <100 cells/sec. The laser excitation is provided at 2 wavelengths of 488 nm supplied by a solid blue state laser at 20mW and 640 nm powered by 14.7mW diode red laser. Green fluorescence (480-530 nm) is measured in the FL-1 channel and red fluorescence (640 nm) in the FL-2 channel. The percentage of positive cells (TUNEL-positive) will be calculated using the flow cytometer software.

Proteomic analysis Individual samples collected from each group will be subjected to 65% percoll gradient to specifically remove the white blood cells. Semen samples will be washed with PBS three times. Once the supernatant is removed, spermatozoa will be solubilized in radio-immunoprecipitation assay (RIPA) lysis buffer containing the proteinase inhibitor cocktail. After complete lysis of the spermatozoa, protein concentration will be determined using a bicinchoninic acid (BCA) kit and equal amounts of proteins will be fractionated using SDS-Page 1D gel electrophoresis. Separated bands will be cut from a single Coomassie blue stained 1D gel and analyzed. The bands will be washed, reduced, alkylated, and digested with trypsin. The digests will be separated by capillary column LC-tandem MS and the CID spectra searched against the human reference sequence database.

Functional annotation and enrichment analysis will be performed using publicly available bioinformatics annotation tools and databases such as GO Term Finder, GO Term Mapper, UniProt, Software Tools for Researching Annotations of Proteins (STRAP), Database for Annotation, Visualization and Integrated Discovery (DAVID) (http://david.niaid.nih.gov), and proprietary software package such as IPA (Ingenuity Pathway Analysis) from Ingenuity® Systems, used to obtain consensus-based, comprehensive functional context for the large list of proteins derived from proteomic study. The data will be subjected to STRING (Search Tool for the Retrieval of Interacting Genes/Proteins), a biological database and web resource of known and predicted protein-protein interactions. This will help in identifying critical proteins involved in reproductive function.

Data analysis All the data will be analyzed using the using the MedCalc Software (V. 17.8; MedCalc Software, Ostend, Belgium). Paired t-test will be used if the distribution is normal. Whereas, Wilcoxon signed rank tests will be used for parameters that do not follow normal distribution. For paired T-test comparisons based on 20 samples for each experiment, the power should be least 90% for parameters where a coefficient of variation is no more than 20%.

ELIGIBILITY:
Inclusion Criteria:

• Normal healthy men with normozoospermic semen parameters.

Exclusion Criteria:

* Subjects with a history of smoking
* Chewing tobacco
* Alcohol consumption
* Antioxidant supplementation
* Orchitis, varicocele, tuberculosis, diabetes mellitus, and hypertension
* Viral/bacterial infection in the past 4 weeks
* History of cardiac, neural, or nephrotic disease
* Family history of any genetic disease

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male subjects, normozoospermic healthy donors.
Enrollment: 40 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Sperm concentration | 0 weeks
  Semen analysis will be carried out using LensHooke™X1 PRO semen quality analyzer. Sperm concentration (millions/ mL) will be assessed in both the groups (Qi-shield user group and sham Qi-shield user group).
Sperm concentration | 4 weeks
  Semen analysis will be carried out using LensHooke™X1 PRO semen quality analyzer. Sperm concentration (millions/ mL) will be assessed in both the groups (Qi-shield user group and sham Qi-shield user group).
Sperm concentration | 8 weeks
  Semen analysis will be carried out using LensHooke™X1 PRO semen quality analyzer. Sperm concentration (millions/ mL) will be assessed in both the groups (Qi-shield user group and sham Qi-shield user group).
Total sperm motility | 0 weeks
  Semen analysis will be carried out using LensHooke™X1 PRO semen quality analyzer. Total motility (%) will be assessed in both the groups (Qi-shield user group and sham Qi-shield user group).
Total sperm motility | 4 weeks
  Semen analysis will be carried out using LensHooke™X1 PRO semen quality analyzer. Total motility (%) will be assessed in both the groups (Qi-shield user group and sham Qi-shield user group).
Total sperm motility | 8 weeks
  Semen analysis will be carried out using LensHooke™X1 PRO semen quality analyzer. Total motility (%) will be assessed in both the groups (Qi-shield user group and sham Qi-shield user group).
Progressive motility | 0 weeks
  Semen analysis will be carried out using LensHooke™X1 PRO semen quality analyzer. Progressive motility (%) will be assessed in both the groups (Qi-shield user group and sham Qi-shield user group).
Progressive motility | 4 weeks
  Semen analysis will be carried out using LensHooke™X1 PRO semen quality analyzer. Progressive motility (%) will be assessed in both the groups (Qi-shield user group and sham Qi-shield user group).
Progressive motility | 8 weeks
  Semen analysis will be carried out using LensHooke™X1 PRO semen quality analyzer. Progressive motility (%) will be assessed in both the groups (Qi-shield user group and sham Qi-shield user group).
Sperm morphology | 0 weeks
  Semen analysis will be carried out using LensHooke™X1 PRO semen quality analyzer. Sperm morphology (%) will be assessed in both the groups (Qi-shield user group and sham Qi-shield user group).
Sperm morphology | 4 weeks
  Semen analysis will be carried out using LensHooke™X1 PRO semen quality analyzer. Sperm morphology (%) will be assessed in both the groups (Qi-shield user group and sham Qi-shield user group).
Sperm morphology | 8 weeks
  Semen analysis will be carried out using LensHooke™X1 PRO semen quality analyzer. Sperm morphology (%) will be assessed in both the groups (Qi-shield user group and sham Qi-shield user group).
Seminal oxidative stress | 0 weeks
  ORP is considered as a marker of oxidative stress. Increased levels of oxidative stress is harmful to the spermatozoa. In semen samples ORP is measured using MiOXSYS analyzers. Seminal ORP will be assessed in both the groups (Qi-shield user group and sham Qi-shield user group) to evaluate the change in the seminal oxidative stress due to use of Qi-shield.
Seminal oxidative stress | 4 weeks
  ORP is considered as a marker of oxidative stress. Increased levels of oxidative stress is harmful to the spermatozoa. In semen samples ORP is measured using MiOXSYS analyzers. Seminal ORP will be assessed in both the groups (Qi-shield user group and sham Qi-shield user group) to evaluate the change in the seminal oxidative stress due to use of Qi-shield.
Seminal oxidative stress | 8 weeks
  ORP is considered as a marker of oxidative stress. Increased levels of oxidative stress is harmful to the spermatozoa. In semen samples ORP is measured using MiOXSYS analyzers. Seminal ORP will be assessed in both the groups (Qi-shield user group and sham Qi-shield user group) to evaluate the change in the seminal oxidative stress due to use of Qi-shield.
Sperm DNA damage | 0 weeks
  Sperm DNA integrity is directly correlated with the quality of the spermatozoa. Increased levels of sperm DNA damage has negative impact on pregnancy and live birth rates. Sperm DNA fragmentation (SDF) is measured using TUNEL assay. In the current study levels of SDF before and after the use of Qi-shield will allow us to understand the effect of electromagnetic radiations on DNA integrity of spermatozoa.
Sperm DNA damage | 4 weeks
  Sperm DNA integrity is directly correlated with the quality of the spermatozoa. Increased levels of sperm DNA damage has negative impact on pregnancy and live birth rates. Sperm DNA fragmentation (SDF) is measured using TUNEL assay. In the current study levels of SDF before and after the use of Qi-shield will allow us to understand the effect of electromagnetic radiations on DNA integrity of spermatozoa.
Sperm DNA damage | 8 weeks
  Sperm DNA integrity is directly correlated with the quality of the spermatozoa. Increased levels of sperm DNA damage has negative impact on pregnancy and live birth rates. Sperm DNA fragmentation (SDF) is measured using TUNEL assay. In the current study levels of SDF before and after the use of Qi-shield will allow us to understand the effect of electromagnetic radiations on DNA integrity of spermatozoa.
Sperm proteome | 0 weeks
  In spermatozoa normal expression of fertility associated proteins are essential for fertilization process. Several studies reported that aberrant expression of proteins related to sperm function as capacitation, hyperactivation, acrosome reaction and binging of zona pellucida with ovum in infertile men. Furthermore, electromagnetic radiations can also cause molecular changes. In the present study, proteome profile of the spermatozoa from subjects before and after the use of Qi-shield will provide the information related to the molecular changes at protein level.
Sperm proteome | 4 weeks
  In spermatozoa normal expression of fertility associated proteins are essential for fertilization process. Several studies reported that aberrant expression of proteins related to sperm function as capacitation, hyperactivation, acrosome reaction and binging of zona pellucida with ovum in infertile men. Furthermore, electromagnetic radiations can also cause molecular changes. In the present study, proteome profile of the spermatozoa from subjects before and after the use of Qi-shield will provide the information related to the molecular changes at protein level.
Sperm proteome | 8 weeks
  In spermatozoa normal expression of fertility associated proteins are essential for fertilization process. Several studies reported that aberrant expression of proteins related to sperm function as capacitation, hyperactivation, acrosome reaction and binging of zona pellucida with ovum in infertile men. Furthermore, electromagnetic radiations can also cause molecular changes. In the present study, proteome profile of the spermatozoa from subjects before and after the use of Qi-shield will provide the information related to the molecular changes at protein level.

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Agarwal, PhD, Principal Investigator — American Center for Reproductive Medicine, Cleveland Clinic
Locations (1):
- American Center for Reproductive Medicine, Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agarwal A, Deepinder F, Sharma RK, Ranga G, Li J. Effect of cell phone usage on semen analysis in men attending infertility clinic: an observational study. Fertil Steril. 2008 Jan;89(1):124-8. doi: 10.1016/j.fertnstert.2007.01.166. Epub 2007 May 4. PMID 17482179
- [Background] Agarwal A, Desai NR, Makker K, Varghese A, Mouradi R, Sabanegh E, Sharma R. Effects of radiofrequency electromagnetic waves (RF-EMW) from cellular phones on human ejaculated semen: an in vitro pilot study. Fertil Steril. 2009 Oct;92(4):1318-1325. doi: 10.1016/j.fertnstert.2008.08.022. Epub 2008 Sep 20. PMID 18804757
- [Background] Agarwal A, Henkel R, Huang CC, Lee MS. Automation of human semen analysis using a novel artificial intelligence optical microscopic technology. Andrologia. 2019 Dec;51(11):e13440. doi: 10.1111/and.13440. Epub 2019 Oct 4. PMID 31583732
- [Background] Desai NR, Kesari KK, Agarwal A. Pathophysiology of cell phone radiation: oxidative stress and carcinogenesis with focus on male reproductive system. Reprod Biol Endocrinol. 2009 Oct 22;7:114. doi: 10.1186/1477-7827-7-114. PMID 19849853
- [Background] Kesari KK, Agarwal A, Henkel R. Radiations and male fertility. Reprod Biol Endocrinol. 2018 Dec 9;16(1):118. doi: 10.1186/s12958-018-0431-1. PMID 30445985
- [Background] Kivrak EG, Yurt KK, Kaplan AA, Alkan I, Altun G. Effects of electromagnetic fields exposure on the antioxidant defense system. J Microsc Ultrastruct. 2017 Oct-Dec;5(4):167-176. doi: 10.1016/j.jmau.2017.07.003. Epub 2017 Aug 2. PMID 30023251